CLINICAL TRIAL: NCT00703768
Title: An Open-Label, Phase ll Trial Comparing FACT-P Scores For Subjects Who Are Indicated To Receive Androgen Deprivation Therapy And Have A Doubling In PSA Post Curative Therapy Of Either Less Than Or Greater Than One Year
Brief Title: Quality of Life for Subjects Receiving Androgen Deprivation Therapy and Have a Doubling in PSA of Either Less Than or Greater Than 1 Year
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Urology South Shore Research Inc. (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Dr. Lorne Aaron, Urology South Shore Research Inc.
Other Study IDs: D8664L00006
Record Dates: First submitted 2008-06-19; First posted 2008-06-23 (Estimated); Last update posted 2009-02-17 (Estimated); Status verified 2009-02

CONDITIONS: Prostate Cancer
Keywords: Quality of Life; Androgen Deprivation Therapy; Goserelin
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- A: Patients who have been identified as having a doubling in PSA from nadir of greater than one year
- B: Patients who have been identified as having a doubling in PSA from nadir of less than one year.

SUMMARY:
The purpose of this study is to evaluate if there is a difference in quality of life (as measured by FACT-P) in patients treated with androgen deprivation therapy (ADT) for biochemical failure (PSA recurrence) following surgery or radiation for prostate cancer depending on when ADT is initiated.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Received therapy of curative intent (surgery or radiotherapy)
* Have a rising PSA which has doubled from a nadir value.
* Histologically proven prostate cancer requiring androgen deprivation therapy for at least 12 months
* Written informed consent to participate in the trial.

Exclusion Criteria:

* Known hypersensitivity to Zoladex, Casodex, ar any component of these products
* Prior treatment with LHRH agonist or anti-androgens in the past 12 months
* Any concomitant condition that would make it undesirable, in the physician's opinion, for the subject to participate in the trial or would jeopardize compliance with the protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male subjects aged 18 years or older with histologically-confirmed prostate cancer, showing biochemical failure (defined as a rising PSA) following definitive therapy (surgery or radiation) and indicated to receive hormone therapy.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2006-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Significant difference in FACT-P scores after 12 months between the 2 groups | 12 months

SECONDARY OUTCOMES:
PSA response | 12 months
To evaluate the ease of use of FACT-P to measure Quality of Life | 12 months
QOL, side effect profile and evaluate the safety and tolerability of Androgen Deprivation Therapy | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lorne Aaron, MD, Principal Investigator
Locations (1):
- Urology South Shore Research Inc., Greenfield Park, Quebec, Canada